CLINICAL TRIAL: NCT03228810
Title: ROR1751: Genetic Biomarker Discovery for Metastatic Prostate Cancer
Brief Title: Genetic Biomarker Discovery for Metastatic Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Cheville, PI, Mayo Clinic
Other Study IDs: 16-007522
Record Dates: First submitted 2017-07-23; First posted 2017-07-25 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men >18 years old with metastatic prostate cancer
  Interventions: Other: Blood draw; Procedure: Tissue biopsy

INTERVENTIONS:
Other: Blood draw — (2) 10 mL tubes will be collected
Procedure: Tissue biopsy — Tissue biopsy of metastatic tissue if undergoing clinical care-directed biopsy

SUMMARY:
Biomarkers from circulating cell-free tumor DNA in peripheral blood will identify patients with metastatic prostate cancer diagnosed with C11 choline PET/CT who will benefit from metastasis-directed radiation, ablative therapies, and/or surgery. Tissue and blood will be collected before treatment. If patients receive androgen deprivation, then blood will be collected after neoadjuvant androgen deprivation but before radiation, ablative therapies, or surgery. Subsequent samples will be obtained at 3 months and 6 months following treatment, after which no further patient contact will occur.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18 years old and older.
* Histologically proven diagnosis of prostate cancer.
* Radiographic evidence of non-regional lymph node involvement, pelvic lymph node recurrence, and/or bone metastases.
* Requiring a clinically directed biopsy or resection of tumor at Mayo Clinic Rochester.
* Receiving local therapy for metastatic disease with radiation, ablative therapies, and/or surgery at Mayo Clinic Rochester.
* Willingness to provide blood sample prior to receipt of treatment, as well as after neoadjuvant androgen deprivation therapy and at 3 months and 6 months after radiation, ablation, or surgery.
* Absence of a second active malignancy.
* An understanding of the protocol and its requirements, risks, and discomforts.
* The ability and willingness to sign an informed consent.

Exclusion Criteria:

* Inability on the part of the patient to understand the informed consent or be compliant with the protocol.
* History of a serious or life-threatening allergic reaction to local anesthetics (i.e., lidocaine, xylocaine).

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Men with metastatic prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Detect cell-free tumor DNA in patients with metastatic prostate cancer | prior to treatment
  tissue biopsy
Calculate cell-free tumor DNA in relation to metastasis-directed radiation and androgen deprivation therapy (ADT) | before and immediately after ADT and at 3 months and 6 months after radiation
  blood draw

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials